CLINICAL TRIAL: NCT03072498
Title: Collection of Bone Marrow, Peripheral Blood (PB), Epithelial Tissue, and Saliva Samples From Patients With Myelodysplastic Syndromes (MDS) to Identify MDS-Specific Antigens (MSA) for Use in Cellular Immunotherapy.
Brief Title: Collection of Samples From Patients With MDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PersImmune, Inc (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: 161345
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Myelodysplastic Syndromes(MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We intend to obtain cells from bone marrow, peripheral blood, epithelial tissue, and saliva from patients who are likely to be candidates for MDS treatment in the near future.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to collect information and bone marrow, blood, saliva, cheek cells and skin to be used in the laboratory to assist the sponsor in identifying a new way of treating MDS.

DETAILED DESCRIPTION:
Goals of the study:

The purpose of this study is to collect the blood and marrow samples, and non-involved fibroblasts, that are required to identify the unique, personalized array of mutation-driven neoantigens that are expressed by the subject's MDS cells and to assess the feasibility of immunizing and expanding one or more of the patient's T cells ex vivo for investigation of their use as adoptive cellular immunotherapy.

ELIGIBILITY:
Patients must meet the following initial inclusion criteria:

* Diagnosis or suspected diagnosis of MDS or CCUS
* Age 18 or older

Patient exclusion criteria:

* Currently receiving or within 3 months has received hypomethylating agent(s), lenalidomide, cytotoxic agents, or within the previous 4 weeks corticosteroids > 5 mg prednisone daily or any other immunosuppressants
* Previous allogenic transplant
* Inability to provide consent
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 24 Subjects (patients and donors) will be recruited over a 3-year period. Both male and female subjects will be included and there will be no restrictions based on race or ethnicity.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-12-05 (Estimated); Study Completion 2021-03-05 (Estimated)

PRIMARY OUTCOMES:
Genomics of patients with MDS | 2 years
  To sequence the exome and transcriptome obtained from MDS hematopoietic cells and the exome from non-hematopoietic cells (e.g. fibroblasts).

SECONDARY OUTCOMES:
Identification of patients' MDS-specific variant | 2 years
  To select variants by comparing MDS versus non-MDS cell exome sequences. MDS-specific variant sequences are defined as those that differ between the two and are not common polymorphisms. We will also compare myeloid and lymphoid hematopoietic cells and assess the number of myeloid-specific vs myeloid and lymphoid MDS-related variants
Immunogenic mutant neoantigen peptide selection | 2 years
  To select putative mutation-driven neoantigen-related peptides, which represent the sequences obtained from Aim 2, according to their ability to bind to the patient's MHC using PersImmune's licensed and proprietary algorithms.
Peptide Immunogenicity confirmation and donor T cell stimulation | 2 years
  To test the neoantigen peptides for their in vitro immunogenicity for autologous T lymphocytes.
Peptide immunogenicity confirmation and donor T cell stimulation | 2 years
  To test the potency and specificity of neoantigen peptide-stimulated T cells for the patient's MDS cells that express the defined neoantigens.
Data analysis and interpretation | 2 years
  To create a database summarizing the data obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Bejar, MD, Principal Investigator — UCSD
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - University of California San Diego, La Jolla, California

IPD SHARING:
Plan to Share IPD: Undecided